CLINICAL TRIAL: NCT03125577
Title: Combination CAR-T Therapy of 4SCAR19 Plus 4SCAR20, 22, 38, 70 and 123 Targeting Hematological Malignancies
Brief Title: Combination CAR-T Cell Therapy Targeting Hematological Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17005
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: B-cell Malignancies
Keywords: 4S CAR-T; CD19; CD20; CD22; CD38; CD123; B cell leukemia; B-ALL; CD70; CD30
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4SCAR19 and 4SCAR20/CD22/CD30/CD38/CD70/CD123 (Experimental): Patients who have relapsed and refractory B cell malignancies after chemotherapy will be treated with CD19 and CD20/CD22/CD30/CD38/CD70/CD123-specific gene-engineered T cells.
  Interventions: Biological: 4SCAR19 and 4SCAR22; Biological: 4SCAR19 and 4SCAR38; Biological: 4SCAR19 and 4SCAR20; Biological: 4SCAR19 and 4SCAR123; Biological: 4SCAR19 and 4SCAR70; Biological: 4SCAR19 and 4SCAR30

INTERVENTIONS:
Biological: 4SCAR19 and 4SCAR22 — 4SCAR19 and 4SCAR22
Biological: 4SCAR19 and 4SCAR38 — 4SCAR19 and 4SCAR38
Biological: 4SCAR19 and 4SCAR20 — 4SCAR19 and 4SCAR20
Biological: 4SCAR19 and 4SCAR123 — 4SCAR19 and 4SCAR123
Biological: 4SCAR19 and 4SCAR70 — 4SCAR19 and 4SCAR70
Biological: 4SCAR19 and 4SCAR30 — 4SCAR19 and 4SCAR30

SUMMARY:
The study will evaluate safety and efficacy of a combination of 4th generation chimeric antigen receptor gene-modified T cells targeting CD19 (4SCAR19) and CD20 (4SCAR20), CD22 (4SCAR22), CD30 (4SCAR30), CD38 (4SCAR38), CD70 (4SCAR70) or CD123 (4SCAR123) for patients with B cell malignancies. Clinical response and development of a standardized lentiviral vector and cell production protocol will be investigated. This is a phase I/II trial enrolling patients from multiple clinical centers.

DETAILED DESCRIPTION:
Background:

T cells modified with lentiviral chimeric antigen receptor (CAR) gene have been studied in different clinical settings. Recent successes suggest that increased costimulatory signaling in the CAR design is critical for long term efficacy. Several clinical reports indicate that many patients still relapse and developed CD19-negative cancer cells after CD19 targeted therapy. Thus, to prevent the target escapes and improve the therapeutic effects, CAR gene-modified T cells targeting CD20, CD22, CD30, CD38, CD70 or CD123 are considered to apply together with CD19 CAR-T cells.

Activation of T cell response to high tumor burden may induce a severe response. To increase safety, a novel design using an inducible caspase 9 fusion gene has been incorporated in the CAR gene. A 4th generation CAR lentiviral vector (4SCAR) carrying multiple costimulatory signals for CD28/CD137/CD27 plus an inducible apoptotic caspase 9 gene has been established. This study aims to evaluate the activities of a combination of CAR gene-modified T cells to target cancer cells based on specific CD19/CD20/CD22/CD30/CD38/CD70/CD123 single chain antibody gene designs (4SCAR19/20/22/30/38/70/123).

Objective:

To evaluate safety and efficacy of administrating 4SCAR19, 4SCAR20, 4SCAR22, 4SCAR30, 4SCAR38, 4SCAR70 and 4SCAR123 T cells to patients with mixed CD19 positive and negative B cell malignancies following a cyclophosphamide/fludarabine based conditioning regimen.

Eligibility:

Patients older than 6-month-old with CD19 positive or negative B cell malignancies that have recurred after or refractory to standard therapy and is deemed incurable using standard treatment.

Design:

Participants will be screened based on cancer cell phenotype analyzed using flow cytometry or immunohistochemical staining methods. Peripheral blood mononuclear cells (PBMC) will be obtained through apheresis. On Day -5 to -7, T cells from PBMC will be activated and enriched, which will be followed by 4SCAR19, 4SCAR20, 4SCAR22, 4SCAR30, 4SCAR38, 4SCAR70 and 4SCAR123 lentiviral transduction. The total cell preparation time is approximately 5-7 days. Participants will receive a preparative conditioning regimen comprising cyclophosphamide/fludarabine to prepare their immune system to accommodate the modified CAR T cells. The preparative regimen will depend on the immune condition of patients, which is consistent with standard chemotherapy conditioning regimen. Participants will receive an infusion of the modified 4SCAR19 and 4SCAR20/22/30/38/70/123 T cells and closely followed up for treatment-related responses. Participants will be continuously monitored for CAR T cells and clinical responses in a preset timeline.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 6 months.
2. malignant B cell surface expression of CD19/CD20/CD22/CD30/CD38/CD70/CD123 molecules.
3. the KPS score over 80 points, and survival time is more than 1 month.
4. greater than Hgb 80 g/L.
5. no contraindications to blood cell collection.

Exclusion Criteria:

1. accompanied with other active diseases, the treatment is difficult to assess patient response.
2. bacteria, fungus, or virus infection, unable to control.
3. living with HIV.
4. active HBV and HCV infection.
5. pregnant and nursing mothers.
6. under systemic steroid treatment within a week of the treatment.
7. prior failed CAR-T treatment.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of fourth generation anti CD19 and CD20/CD22/CD30/CD38/CD70/CD123 CAR-T cells in patients with relapsed B cell malignancies using CTCAE 4 standard to evaluate the level of adverse events standard to evaluate the level of adverse events | 24 weeks
  physiological parameter (for safety, measuring cytokine response, fever, symptoms)

SECONDARY OUTCOMES:
Anti tumor activity of fourth generation anti CD19 and CD20/CD22/CD30/CD38/CD70/CD123 CAR-T cells in patients with relapsed or refractory B cell malignancies | 1 year
  scale of CAR copies and leukemic cell burden (for efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (3):
- China (3):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nair S, Wang JB, Tsao ST, Liu Y, Zhu W, Slayton WB, Moreb JS, Dong L, Chang LJ. Functional Improvement of Chimeric Antigen Receptor Through Intrinsic Interleukin-15Ralpha Signaling. Curr Gene Ther. 2019;19(1):40-53. doi: 10.2174/1566523218666181116093857. PMID 30444200